CLINICAL TRIAL: NCT06045702
Title: Establishment of a Primary Epididymal Cell Model From Epididymal Samples to Study CFTR Gene Regulation
Acronym: CFTR-EP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0273
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Cystic Fibrosis; Congenital Bilateral Absence of Vas Deferens; Sterility, Male
Keywords: Infertility; Primary epididymal cells
MeSH Terms: conditions — Cystic Fibrosis; Congenital bilateral aplasia of vas deferens; Infertility, Male; Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group control: Adult patients with no genetic pathology other than male infertility of any type leading to an inability to procreate without medical assistance, and requiring surgery to recover spermatozoa for possible in vitro fertilization.
  Interventions: Procedure: Epididymal sample
- CFTR-associated pathology: Major patients with cystic fibrosis or male infertility due to agenesis of the vas deferens. These patients will be included in the study because they have the prospect of procreation by in vitro fertilisation requiring surgery to recover spermatozoa.
  Interventions: Procedure: Epididymal sample

INTERVENTIONS:
Procedure: Epididymal sample — During a planned surgical procedure carried out by the Urology and Medically Assisted Reproduction (MAP) department at Brest University Hospital in the patients included in the study, a remnant epididymal sample (between ½ and ¼ of a cc) will be kept for research purposes. These patients suffer from male infertility, leading them to undergo surgery in order to check for the presence of spermatozoa in the epididymis, and to recover spermatozoa which will be frozen and flaked in the AMP department of the CHU Brest, in the event of future procreation by in vitro fertilisation.

SUMMARY:
The aim of this observational study is to better understand the role and involvement of the regulatory elements of the CFTR gene, with the aim of better describing the 3D organisation of chromatin at the CFTR locus in epididymal cells in patients with male infertility of any kind, or with cystic fibrosis or bilateral agenesis of the vas deferens, requiring scheduled surgery.

The main questions it aims to answer are:

* to better characterise this 3D organisation of the CFTR locus, the study of regulatory elements in primary epididymal cells is the most relevant and realistic model.
* to gain a better understanding of the regulation of the CFTR gene in epididymal cells in order to gain a better understanding of the pathology of male infertility caused by bilateral agenesis of the vas deferens, a symptom and also a borderline form of cystic fibrosis.

Participants will Epididymal samples will be taken by a urologist for the AMP department during the planned surgery. The rest of the samples taken will be recovered for research purposes, with the aim of recovering the epididymal cells contained in the sample. This is in no way an additional procedure and will have no impact on the patient's health..

ELIGIBILITY:
Inclusion Criteria:

* Male patients over 18 years of age
* Patients, without genetic pathology, scheduled for epididymal sampling surgery
* Patients with cystic fibrosis or bilateral vas deferens agenesis, scheduled for epididymal sampling surgery.
* Signature of a consent form

Exclusion Criteria:

* Patients not scheduled for epididymal harvesting surgery
* Patients under legal protection (guardianship, curatorship)
* Refusal to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population for this study will be adult male patients with all types of male infertility due to genital defects, including epididymal defects due to obstruction or agenesis of the vas deferens, cystic fibrosis or male infertility due to bilateral agenesis of the vas deferens.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
3D organisation of chromatin at the CFTR locus | 2 years
  Cultur Cell Model

CONTACTS AND LOCATIONS:
Overall Officials: Antoine VALERI, MD,PhD, Principal Investigator — University Hospital, Brest
Locations (1):
- Antoine VALERI, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.